CLINICAL TRIAL: NCT00004667
Title: Phase I Study of Human Von Willebrand Factor for Von Willebrand's Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Center for Research Resources (NCRR) (NIH)
Collaborators: University of North Carolina (Other)
Organization: Office of Rare Diseases (ORD) (NIH)
Purpose: Treatment
Other Study IDs: 199/11955; UNCCH-826
Record Dates: First submitted 2000-02-24; First posted 2000-02-25 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2001-12

CONDITIONS: Von Willebrand's Disease
Keywords: hematologic disorders; rare disease; von Willebrand's disease
MeSH Terms: conditions — von Willebrand Diseases; Hematologic Diseases; Rare Diseases | interventions — von Willebrand Factor

INTERVENTIONS:
Drug: von Willebrand factor

SUMMARY:
OBJECTIVES: I. Evaluate the effect of a new von Willebrand factor concentrate on bleeding time, in vivo recovery, and circulating half-life of the infused factor in patients with von Willebrand's disease.

II. Assess the safety of von Willebrand factor in these patients.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: Patients receive 1 dose of von Willebrand factor concentrate. Timed blood studies are performed for the next 96 hours.

Patients are followed every 2 weeks for 16 weeks, and at 24, 36, and 52 weeks.

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

* von Willebrand's disease

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10
Dates: Start 1993-10

CONTACTS AND LOCATIONS:
Overall Officials: Gilbert C. White, Study Chair — University of North Carolina

REFERENCES:
- [Background] Menache D, Aronson DL, Darr F, Montgomery RR, Gill JC, Kessler CM, Lusher JM, Phatak PD, Shapiro AD, Thompson AR, White GC 2nd. Pharmacokinetics of von Willebrand factor and factor VIIIC in patients with severe von Willebrand disease (type 3 VWD): estimation of the rate of factor VIIIC synthesis. Cooperative Study Groups. Br J Haematol. 1996 Sep;94(4):740-5. doi: 10.1046/j.1365-2141.1996.d01-1860.x. PMID 8826903